CLINICAL TRIAL: NCT02625662
Title: Facioscapulohumeral Dystrophy in Children: a Prospective, Observational Study on the Natural History, Predictors and Clinical Impact (iFocus)
Brief Title: Facioscapulohumeral Dystrophy in Children
Acronym: iFocus
Status: Completed | Type: Observational
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Leiden University Medical Center (Other); Princess Beatrix Muscle Foundation (Other)
Responsible Party: Principal Investigator, RJM Goselink, Prof. dr. Baziel van Engelen, University Medical Center Nijmegen
Other Study IDs: NL53213.091.15
Record Dates: First submitted 2015-12-02; First posted 2015-12-09 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Neurological Observations; Facioscapulohumeral Muscular Dystrophy; Pediatric Disorder
Keywords: muscular dystrophy; natural history; genetic profilling
MeSH Terms: conditions — Neurologic Manifestations; Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- iFSHD group: First recruitment group

SUMMARY:
This study will focus on the symptoms, natural history and clinical impact of facioscapulohumeral muscular dystrophy (FSHD) in children.

Symptoms of classical FSHD start in adulthood. However, a small subgroup of FSHD patients have an early, childhood onset. This early onset is associated with faster progression and other symptoms like hearing loss and epilepsy.

The symptoms, natural history and clinical impact of FSHD in children are largely unknown.

The results of this study will be vital for adequate symptomatic management and trial-readiness.

DETAILED DESCRIPTION:
FSHD is a hereditary muscle disease with slowly progressive muscle weakness. In children it is a very heterogenic disease ranging from severely affected infants to mildly affected adolescents. Symptoms can include muscle weakness, pain, fatigue, epilepsy, hearing loss, vision loss, mental retardation and spinal deformities. The prevalence of these symptoms and the adequate follow-up of these symptoms is unknown. Moreover the clinical impact and social functioning of children with FSHD is under exposed.

Therefore this study will focus on the total spectrum of FSHD in children.

In addition, an extensive genetic screening will be conducted, searching for (epi)genetic disease modifiers and severity predictors.

ELIGIBILITY:
Inclusion Criteria:

* aged 0-17 years
* symptoms of facial, scapulohumeral or peroneal weakness
* genetically proven FSHD1 or FSHD2
* living in the Netherlands

Exclusion Criteria:

* no informed consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children aged 0-17 years with genetically confirmed FSHD
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Motor Function Measure | 2 years
  Global motor functioning

SECONDARY OUTCOMES:
ICH Body functioning: Manual Muscle Testing | 2 years
  Manual Muscle Testing using the 5-point scale of the Medical Research Council.
ICH Body functioning: 6 Minute Walk test | 2 years
  Walking Distance in 6 minutes.
ICH Body functioning: Denver II developmental screening test | 2 years
  Developmental level.
ICH Body functioning: visual acuity | 2 years
  Snellen card
ICH Body functioning: hearing | 2 years
  Tone- and voice audiometry
ICH Body functioning: mental functioning | 2 years
  Electro-encephalography performed in clinically suspected epilepsy.
ICH Body functioning: Pain | 2 years
  Faces scale pain.
ICH Body functioning: cardiac functioning | 2 years
  12 lead Electrocardiogram.
ICH Body functioning: respiratory functioning | 2 years
  Upright sitting spirometry measuring vital capacity and forced expiratory volume.
ICH Body functioning: muscle functions | 2 years
  FSHD-evaluation score, Ricci score.
ICH Body functioning: ingestion functions | 2 years
  TOMASS-C test.Neuromuscular disease swallowing status scale.
ICH Body structure: muscle ultrasonography | 2 years
  Quantitative muscle ultrasonography of 20 skeletal muscles.
ICH Body structure: eye structure | 2 years
  Dilated fundoscopy, optical coherence tomography, slit lamp examination
ICF: Activities and participation: Kidscreen | 2 years
  Kidscreen-52.
ICF: Activities and participation: NeuroQol | 2 years
  NeuroQol fatigue domain, qualitative anamnesis.
ICF: Activities and participation: SEV | 2 years
  SEV questionnaire: social-emotional functioning.
(Epi)genetic disease-modifying factors | 2 years
  Genetic profiling (DNA and RNA).
Prevalance estimation | 2 years
  Nationwide recruitment, prevalence estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Baziel van Engelen, MD, PhD, Principal Investigator — Nijmegen University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Patients have not given consent for IPD. Please contact researchers.

REFERENCES:
- [Derived] Goselink RJ, Schreuder TH, Mul K, Voermans NC, Pelsma M, de Groot IJ, van Alfen N, Franck B, Theelen T, Lemmers RJ, Mah JK, van der Maarel SM, van Engelen BG, Erasmus CE. Facioscapulohumeral dystrophy in children: design of a prospective, observational study on natural history, predictors and clinical impact (iFocus FSHD). BMC Neurol. 2016 Aug 17;16:138. doi: 10.1186/s12883-016-0664-6. PMID 27530735